CLINICAL TRIAL: NCT01791946
Title: Binocular Treatment of Amblyopia Before and After Strabismus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-186H
Record Dates: First submitted 2013-02-07; First posted 2013-02-15 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2015-10

CONDITIONS: Amblyopia; Strabismus
Keywords: lazy eye; cross eye; cross eyed
MeSH Terms: conditions — Amblyopia; Strabismus; Esotropia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment Group A (Post-Surgery) (Experimental): Subjects enrolled in this arm will first have eye alignment corrective surgery and then complete six weeks of the investigational binocular treatment training.
  Interventions: Procedure: Binocular Treatment
- Treatment Group B (Pre-Surgery) (Experimental): Subjects enrolled in this arm will first complete six weeks of the investigational binocular treatment training and then have eye alignment corrective surgery.
  Interventions: Procedure: Binocular Treatment
- Sham Treatment (Sham Comparator): Subjects enrolled in this arm will first complete six weeks of the sham binocular treatment and then undergo eye alignment corrective surgery.
  Interventions: Procedure: Sham Binocular Treatment

INTERVENTIONS:
Procedure: Binocular Treatment — The binocular treatment involves the completion of visual tasks via virtual reality goggles. The stimulus is presented to each eye separately, allowing for varying levels of contrast to be presented to each eye. (The visual task is therefore made more or less difficult with the variation of contrast presented to either eye.) Subjects will complete the computer-based visual tasks for approximately 36 hours total over the course of six weeks, or six hours per week for six weeks.
  Arms: Treatment Group A (Post-Surgery); Treatment Group B (Pre-Surgery)
Procedure: Sham Binocular Treatment — The sham treatment involves the same computer-based visual tasks and timeframe as the binocular treatment training but there will be no variation in contrast presentation to either eye.
  Arms: Sham Treatment

SUMMARY:
The primary objective of this study is to assess the effectiveness of an investigational binocular treatment in improving vision in strabismic amblyopes (i.e., patients with lazy eye, or poor vision in one eye due to a present or former eye misalignment). Patients will be randomized to receive the study treatment either before or after strabismus surgery (i.e., corrective eye alignment surgery) or sham treatment before surgery. The study hypothesis is that there will be no significant change in vision in neither the pre nor post-surgery groups and no significant change in vision in neither the sham nor actual treatment groups.

DETAILED DESCRIPTION:
This is a placebo-controlled, partially-randomized clinical trial. The patients will be assigned to one of two groups, Treatment Group A or Treatment B group. To help minimize bias, a blinded staff member will perform the visual acuity assessments throughout the study. The PI and Sub-I's will remain blinded to the treatment groups so that they may perform the visual exams throughout the study, if necessary.

Patients who have had strabismus surgery prior to being recruited will be allowed to participate in the study and, if eligible, will be automatically assigned to Treatment Group A.

Patients who are scheduled to have strabismus surgery at least six weeks from their screening clinic visit will be allowed to participate, once eligibility is determined. These patients will be included in Treatment Group B and randomized to either actual treatment or sham treatment. Each eligible participant will be included in the study and blinded as to which treatment group s/he has been assigned.

The duration of each subject's participation in the study will be about 7.5 months. All subjects will have a baseline visit to assess eligibility. Subjects in Treatment Group A will undergo strabismus surgery, if it was not previously performed, followed by 6 weeks of binocular treatment and a 3-6 month follow-up period. NOTE: There will be 4-6 weeks between surgery and the start of treatment to allow for full post-surgery recovery before starting treatment. Subjects in Treatment Group B will undergo 6 weeks of treatment/sham followed by strabismus surgery and a 3-6 month follow-up period.

If a treatment effect on vision is found, participants enrolled in the sham treatment arm will be offered the binocular treatment at the conclusion of the study and following surgery. Sham participants will be allowed to receive the study treatment so long as they have completed the study and there is no presence of any new medical condition following surgery that would be considered reasons for exclusion by the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Presence of amblyopia in one eye due to congenital strabismus.
* Amblyopic eye has a fully-corrected visual acuity of 20/30 or less with no other cause for the visual loss except amblyopia.
* Patient is 18 to 60 years old.
* Corrected vision in other eye is normal.
* Eligible for strabismus surgery or has completed it previously with a successful outcome, as determined by the treating physician.
* Available and willing to comply with examination procedures and schedule.
* Signed and dated informed consent.

Exclusion Criteria:

* Fully-corrected visual acuity of less than 20/30 in both eyes.
* Visual decrement due to anything other than amblyopia.
* At high risk for developing intractable diplopia (double vision) if vision in weak eye is improved. (To be determined by treating physician.)
* Unable or unavailable to complete at least 18 hours of binocular treatment over the course of six weeks.
* Currently enrolled in another research study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2013-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome variable is a composite of the difference in visual acuity and stereo vision measurements taken before binocular treatment and strabismus surgery versus after binocular treatment and strabismus surgery. | This is a change outcome measure. That is measurements will be taken at baseline, 6 weeks, and approximately 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Dean Cestari, M.D., Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
We do not [plan on sharing IPD with other researchers.

REFERENCES:
- [Result] Hess RF, Mansouri B, Thompson B. Restoration of binocular vision in amblyopia. Strabismus. 2011 Sep;19(3):110-8. doi: 10.3109/09273972.2011.600418. PMID 21870914
- [Result] Hess RF, Mansouri B, Thompson B. A new binocular approach to the treatment of amblyopia in adults well beyond the critical period of visual development. Restor Neurol Neurosci. 2010;28(6):793-802. doi: 10.3233/RNN-2010-0550. PMID 21209494